CLINICAL TRIAL: NCT00536432
Title: Early Re-intervention in Infants and Small Children After Correction of Tetralogy of Fallot: Prospective Analysis of Myocardial Benefit Using Cardiac MRI and Echocardiography
Brief Title: Early Re-intervention in Infants and Small Children After Correction of Tetralogy of Fallot
Status: Completed | Type: Observational
Sponsor: Competence Network for Congenital Heart Defects (Other Government)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Other Study IDs: MP 4.2
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2010-10

CONDITIONS: Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Tetralogy of Fallot is one of the most frequent congenital heart malformations. In many cases re-interventions, surgical or catheter-based, are necessary after the repair of tetralogy of Fallot in infancy. At present, informations in the literature about the myocardial benefit and the timing of re-interventions are missing in this age group. On the other hand, Fallot patients are dependent on solid criteria for re-interventions, because further interventions like replacement of the pulmonary valve or balloon dilatations of peripheral pulmonary stenoses are common.

The objective of this study is to assess the benefit of such interventions for the right ventricular function. By performing extensive standardised examinations (including MRI, echocardiography, tissue Doppler,,3D-echocardiography, holter monitoring and quality of life assessments) before and 6 to 9 months after the re-intervention data of the right ventricular function are collected. Based on these quantitative data predictive parameters concerning the right ventricular recovery and information about the time of re-intervention should be determined.

DETAILED DESCRIPTION:
In the repair of tetralogy of Fallot, pulmonary insufficiency used to be tacitly accepted as a result of extensive transannular patching (TAP) and considered unobjectionable. In fact, this is well tolerated during the first postoperative years, but today there is increasing evidence that the resulting chronic volume stress to the right ventricle is harmful on the long run, in particular if there are stenoses of the pulmonary artery in addition. Such stenoses, partly due to distortions after shunt surgery, together with pulmonary insufficiency, lead to a combined volume and pressure load of the right ventricle. The chronic volume stress results in a decrease in biventricular function and exercise tolerance, associated with increasing electrical instability with frequent, mostly ventricular, dysrhythmias. This constellation brings about a significantly increased risk of cardiac death.

Pulmonary valve replacement can improve haemodynamics, exercise tolerance and dysrhythmia. However, it is still unclear, which criteria best indicate the need for re-intervention, such as balloon dilatations of peripheral pulmonary stenoses, and what may be the best point in time in infancy.

The objective of this study is to assess the effectiveness of such interventions to the right ventricular function in small children. The data obtained are supposed to determine predictive parameters of the right ventricular recovery and to help to establish criteria for the necessity and time of re-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient's legal representatives
* Patients with tetralogy of Fallot (including pulmonary atresia with vsd) after corrective operation
* Patients < 8 years with corrective surgery and necessary re-intervention (e.g.cardiac catheter intervention or re-operation )

Exclusion Criteria:

* DORV (if there is another VSD than subaortic)
* Associated severe heart defects (e. g. AV canal)
* Other clinically relevant diseases, such as malignant tumor (in the investigating physician's assessment)
* MRI contraindication, e.g. cardiac pacemaker, implanted neurostimulators and other magnetizable foreign bodies

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children, <8 years, with tetralogy of Fallot
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Sarikouch, MD, Principal Investigator — Medizinische Hochschule Hannover, Lower Saxony; Philipp Beerbaum, MD, Study Chair — Evelina Children's Hospital, Guy's and St. Thomas Foundation Trust, Interdisciplinary Medical Imaging Group, King's College London
Locations (14):
- Germany (14):
  - Universitätsklinikum Freiburg, Klinik III Päd. Kardiologie, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Tuebingen, Klinik für Kinderheilkunde und Jugendmedizin, Tübingen, Baden-Wurttemberg
  - Deutsches Herzzentrum Muenchen, Munich, Bavaria
  - Medizinische Hochschule Hannover, Pädiatrische Kardiologie und Intensivmedizin, Hanover, Lower Saxony
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, North Rhine-Westphalia
  - Herzzentrum Duisburg, Kinderkardiologie, Duisburg, North Rhine-Westphalia
  - Universitätsklinikum Essen, Klinik für Kinderkardiologie, Essen, North Rhine-Westphalia
  - Universitätsklinikum Muenster, Klinik für Kinderkardiologie, Münster, North Rhine-Westphalia
  - Deutsches Kinderherzzentrum St. Augustin, Sankt Augustin, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Klinik für Pädiatrische Kardiologie, Homburg/Saar, Saarland
  - Herzzentrum Leipzig, Klinik für Kinderkardiologie, Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Klinik für Kinderkardiologie, Kiel, Schleswig-Holstein
  - Deutsches Herzzentrum Berlin, Berlin, State of Berlin
  - Universitätsklinikum Charite, Campus Virchow-Klinikum, Otto-Heubner-Centrum für Kinder- und Jugendmedizin, Berlin, State of Berlin

REFERENCES:
- See also: click here for more information about the Competence Network for Congenital Heart Defects — http://www.kompetenznetz-ahf.de